CLINICAL TRIAL: NCT03102398
Title: An Open-Label Phase I/IIa Study to Assess the Safety and Tolerability Profile of TR399 in Healthy Volunteers and Erectile Dysfunction Patients
Brief Title: A Study to Assess the Safety and Tolerability Profile of TR399 in Healthy Volunteers and Erectile Dysfunction Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tritech Biopharmaceuticals Co., Ltd. (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR399
Record Dates: First submitted 2017-03-20; First posted 2017-04-05 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; PDE5 inhibitor; Sexual Dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological | interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm and Open-label Study (Experimental)
  Interventions: Drug: TR-399 (5% Vardenafil HCl·3H2O, topical gel)

INTERVENTIONS:
Drug: TR-399 (5% Vardenafil HCl·3H2O, topical gel) — 5% Vardenafil HCl·3H2O, topical gel, 2 drops (50ul, 2.5mg), q.d.

SUMMARY:
The purpose of this phase I/IIa study is to assess the safety and tolerability profile of TR399 in healthy volunteers and erectile dysfunction patients. This study will be conducted via a single-arm and open-label fashion.

DETAILED DESCRIPTION:
Several oral medications containing PDE5 inhibitors, including sildenafil (Viagra®, Pfizer), vardenafil (Levitra®, Bayer) and tadalafil (Cialis®, Lilly), have been marketed for the treatment of ED. Many considerations should be taken before patients are prescribed with PDE5 inhibitor medications, which may cause systemic side effects and should not be taken with nitrates or alpha-blockers.

The active pharmaceutical ingredient (API) of TR399 is 5% Vardenafil HCl·3H2O. Non-clinical studies have shown that the topical use of TR399 can enhance erection and sexual behavior in animal models without causing irritancy and phototoxicity.

This study is designed as a single-arm and open-label fashion in order to explore the safety and PK of TR399 in healthy volunteers, as well as the safety, PK and efficacy of TR399 in patients with ED.

ELIGIBILITY:
Inclusion Criteria:

* Phase I

  1. Male aged between 20~40 years old ;
  2. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, and electrocardiogram;
  3. Body mass index (BMI) between 18.5 and 27, inclusive, (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2]);
  4. Clinically normal, including non-clinical significant abnormal, hematology, biochemistry and urinalysis determinations based on investigator's discretion;
  5. Subject is willing and able to comply with study procedures and has signed informed consent.
  6. With Erectile Function domain of the IIEF score of 25~30
* Phase IIa

  1. Male aged between 20~70 years old ;
  2. Diagnosed and confirmed ED for at least 6 months, defined as "the inability to achieve and maintain an erection of the penis sufficient to complete satisfactory sexual intercourse" by the National Institutes of Health (NIH) consensus report 1993;
  3. With Erectile Function domain of the IIEF score of 13~24;
  4. Stable relationship for more than 3 months;
  5. At least 4 sexual intercourse attempts at 4 different days during 4-week period prior the screening;
  6. With a testosterone level ≥ 240 ng/dL (either naturally or through androgen replacement therapy);
  7. Subject is willing and able to comply with study procedures and has signed informed consent.

Exclusion Criteria:

* Phase I

  1. Known or suspected allergy, hypersensitivity, or intolerance to any ingredients of study product
  2. Subject who has a history or evidence of a medical condition that would expose him to an undue risk of a significant adverse event or interfere with the assessments of safety or pharmacodynamics variables during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, musculoskeletal or hematological disease as determined by the clinical judgment of the investigator
  3. Subject has received any investigational agent within 4 weeks prior to the screening visit
  4. Subject has taken or potentially takes any prescription medication and/or over-the-counter medication from 1 week prior to the screening visit to the end of treatment (Day 15)
  5. Sexual partner is a pregnant or lactating female or a female with childbearing potential not taking reliable contraceptive methods during study period Note: Acceptable contraceptive forms include

     1. Established use of oral, injected or implanted hormonal methods of contraception
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
     3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
  6. Use of PDE-5 inhibitors within the last 2 weeks prior to the screening visit
  7. Use of alpha blockers or nitrates within 2 weeks prior to the screening visit
  8. Subject who has prolongation of QT interval >500 ms (long QT syndrome)
  9. Any of the following hematologic abnormalities:

     1. Hemoglobin < 10.0 g/dL
     2. ANC < 1,500/μL,
     3. Platelets < 75,000 /μL
  10. Any of the following serum chemistry abnormalities:

      1. Total bilirubin > 1.5 × ULN,
      2. gamma-GT > 2.5 x ULN,
      3. Alk-P > 2.5 x ULN,
      4. Serum albumin < 3.0 g/dL, e Any other ≥ Grade 2 laboratory abnormality (based on CTCAE) at Screening visit (other than those listed above)
  11. With history of stroke, myocardial infarction, or Coronary Artery Bypass Graft (CABG) surgery within the last 6 months prior to the screening visit
  12. With history of cardiac failure (NYHA class 2 or above), unstable angina, or life-threatening arrhythmia within the last 6 months prior to the screening visit Note: NYHA = New York Heart Association
  13. With blood pressures as systolic blood pressure <90mmHg or > 170mmHg or diastolic blood pressure <50mmHg or > 120 mmHg
  14. History of orthostatic hypotension Note: Orthostatic hypotension is defined as a decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg.
  15. History of syncope
  16. Hereditary degenerative retinal disorders
  17. History of loss of vision because of NAION (Non-arteritic anterior ischemic optic neuropathy), temporary or permanent loss of vision
  18. Skin diseases, infection or cuts in penile area
  19. History of psychiatric disorder
  20. History of spinal cord injury
  21. Use of HIV protease inhibitors (strong cytochrome P450 CYP3A4 inhibitors), such as indinavir or ritonavir within 2 weeks prior to the screening visit
  22. History of left ventricular outflow obstruction, such as aortic stenosis and hypertrophic cardiomyopathy
  23. With any cardiovascular disorder that is not suitable for sexual activities.
  24. Use of antiarrhythmic agents class IA (such as quinidine, or procainamide) and class III (such as amiodarone or sotalol) within 2 weeks prior to the screening visit
  25. With priapism, such as sickle cell anemia, multiple myeloma or leukemia
* Phase IIa

  1. Known or suspected allergy, hypersensitivity, or intolerance to any ingredients of study product
  2. Participated in another clinical trial and received any investigational drug within four weeks prior to the screening visit
  3. Impaired hepatic function defined as alanine aminotransferase/aspartate aminotransferase (ALT/AST) or alkaline phosphatase (ALP) at least 2.5 times upper referenced limit
  4. Impaired renal function defined as serum-creatinine at least 1.3 mg/dL (at least 115 mmol/L)
  5. With history of stroke, myocardial infarction, or Coronary Artery Bypass Graft (CABG) surgery within the last 6 months prior to the screening visit
  6. With history of cardiac failure (NYHA class 2 or above), unstable angina, or life-threatening arrhythmia within the last 6 months prior to the screening visit Note: NYHA = New York Heart Association
  7. With blood pressures as systolic blood pressure <90mmHg or > 170mmHg or diastolic blood pressure <50mmHg or > 120 mmHg
  8. With any uncontrolled illness or a history of any illness judged by the investigator that entering the trial may be detrimental to the patient
  9. Current treatment with systemic corticosteroids
  10. History of prostatectomy due to prostate cancer, including nerve-sparing techniques
  11. Use of alpha blockers or nitrates within 4 weeks prior to the screening visit
  12. Use of PDE-5 inhibitor, or other treatments for erectile dysfunction within the last 4 weeks prior to the screening visit
  13. Sexual partner is a pregnant or lactating female or a female with childbearing potential not taking reliable contraceptive methods during study period Note: Acceptable contraceptive forms include

      1. Established use of oral, injected or implanted hormonal methods of contraception
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
  14. ED due to structural abnormality of the penis
  15. With a history of HIV infection Note: HIV = Human Immunodeficiency Virus
  16. Subject who has prolongation of QT interval >500 ms (long QT syndrome)
  17. Any of the following hematologic abnormalities:

      1. Hemoglobin < 10.0 g/dL
      2. ANC < 1,500/μL,
      3. Platelets < 75,000 /μL
  18. Any of the following serum chemistry abnormalities:

      1. Total bilirubin > 1.5 × ULN,
      2. gamma-GT > 2.5 x ULN,
      3. Alk-P > 2.5 x ULN,
      4. Serum albumin < 3.0 g/dL, e Any other ≥ Grade 2 laboratory abnormality (based on CTCAE) at Screening visit (other than those listed above)
  19. History of orthostatic hypotension Note: Orthostatic hypotension is defined as a decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg
  20. History of syncope
  21. Hereditary degenerative retinal disorders
  22. History of loss of vision because of NAION (Non-arteritic anterior ischemic optic neuropathy), temporary or permanent loss of vision
  23. Skin diseases, infection or cuts in penile area
  24. History of psychiatric disorder
  25. History of spinal cord injury
  26. Use of HIV protease inhibitors (strong cytochrome P450 CYP3A4 inhibitors), such as indinavir or ritonavir, within 2 weeks prior to the screening visit
  27. History of left ventricular outflow obstruction, such as aortic stenosis and hypertrophic cardiomyopathy
  28. With any cardiovascular disorder that is not suitable for sexual activities.
  29. Use of antiarrhythmic agents class IA (such as quinidine, or procainamide) and class III (such as amiodarone or sotalol), within 2 weeks prior to the screening visit
  30. With priapism, such as sickle cell anemia, multiple myeloma or leukemia

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Diagnosed and confirmed ED for at least 6 months, defined as "the inability to achieve and maintain an erection of the penis sufficient to complete satisfactory sexual intercourse" by the National Institutes of Health (NIH) consensus report 1993
Enrollment: 26 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of TR399 assessed by Incidence of AEs and SAEs | 24 days
  Phase I Incidence of AEs and SAEs
Safety and efficacy evaluation of TR399 assessed by change from baseline to the last evaluation visit during the treatment period in score of IIEF-15 Erectile Function domain | 83 days
  Phase IIa Change from baseline to the last evaluation visit during the treatment period in score of IIEF-15 Erectile Function domain

SECONDARY OUTCOMES:
Safety evaluation of TR399 assessed by Maximum Plasma Concentration (Cmax) | 24 days
  PK profiles - Maximum Plasma Concentration (Cmax) will be measured for safety evaluation of TR399 of Phase I
Safety evaluation of TR399 assessed by Area Under the Curve (AUC) | 24 days
  PK profiles - Area Under the Curve (AUC) will be measured for safety evaluation of TR399 of Phase I
Safety evaluation of TR399 assessed by Time of maximum concentration (Tmax) | 24 days
  PK profiles - Time of maximum concentration (Tmax) will be measured for safety evaluation of TR399 of Phase I
Change from baseline to post-treatment visits in score of IIEF-15 Erectile Function domain | 83 days
  Score of IIEF-15 Erectile Function will be assessed for efficacy evaluation of TR399 of Phase IIa
Change from baseline to post-treatment visits in SEP Question 2 | 83 days
  SEP Question 2 will be assessed for efficacy evaluation of TR399 of Phase IIa
Change from baseline to post-treatment visits in SEP Question 3 | 83 days
  SEP Question 3 will be assessed for efficacy evaluation of TR399 of Phase IIa
Changes from baseline to post-treatment visits in vital signs, physical examination and laboratory examination results | 83 days
  Vital signs, physical examination and laboratory examination results will be assessed for safety evaluation of TR399 of Phase IIa
Incidence of AEs and SAEs | 83 days
  Incidence of AEs and SAEs will be assessed for safety evaluation of TR399 of Phase IIa
Safety evaluation of TR399 assessed by Maximum Plasma Concentration (Cmax) for the first 6 evaluable ED patients | 45 days
  PK profiles - Maximum Plasma Concentration (Cmax) will be measured for safety evaluation of TR399 of Phase IIa
Safety evaluation of TR399 assessed by Area Under the Curve (AUC) for the first 6 evaluable ED patients | 45 days
  PK profiles - Area Under the Curve (AUC) will be measured for safety evaluation of TR399 of Phase IIa
Safety evaluation of TR399 assessed by Time of maximum concentration (Tmax) for the first 6 evaluable ED patients | 45 days
  PK profiles - Time of maximum concentration (Tmax) will be measured for safety evaluation of TR399 of Phase IIa

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No